CLINICAL TRIAL: NCT02130401
Title: Examining the Effects of Neuromodulation on Glucose Metabolism in Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment (15 planned, only 6 enrolled)
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNS-DIA-01
Record Dates: First submitted 2014-04-30; First posted 2014-05-05 (Estimated); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: neuromodulation; caloric vestibular stimulation; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caloric Vestibular Stimulation (CVS) (Experimental): The TNM Device will provide a standardized active thermal waveform that will be used for all patients. The device is non-invasive and does not use electrical stimulation.
  Interventions: Device: TNM Device

INTERVENTIONS:
Device: TNM Device — The device is worn like a music headset and the patient lies on a wedge pillow while the device is active. Each session lasts under 20 minutes.

SUMMARY:
This is an open-label, proof of concept study with a single active treatment arm designed to assess whether CVS-based stimulation has a beneficial effect on patients with type 2 diabetes. The primary outcome measure is a difference between pre and post-treatment A1c.

ELIGIBILITY:
Inclusion Criteria

A subject is eligible for the study if all of the following criteria are met:

* Provide written informed consent prior to enrollment.
* Is male or female between 18-70 years old.
* Has been diagnosed with type II diabetes for greater than 12 months.
* Is currently either using lifestyle modification or taking one or two of the following oral antihyperglycemic agents and has been on stable doses for 90 days prior to screening:

  * metformin
  * DPP-4 inhibitors (sitagliptin, saxagliptin, alogliptin, linaglyptin)
  * Pioglitazone
* Has an A l c between 7.5 - 9.0% based upon point of care testing performed at visit 1.
* Currently performs self-monitoring blood glucose checks at least 3 times per week.
* Able to adhere to protocol requirements.

Exclusion Criteria

A subject will be excluded if any of the following criteria are met:

* Has Type 1 Diabetes or Gestational Diabetes.
* Is pregnant or planning to become pregnant during the course of the study.
* Current use OR use in the past 6 months of sulfonylureas.
* Current use OR use in the past 6 months of insulin
* History of cardiovascular disease or cerebrovascular disease.
* Any planned surgery during the course of the study.
* Current continuous renal replacement therapy.
* Current oral or injectable steroid use or use within the previous 3 months.
* Previous or current treatment with deep brain stimulation.
* Any previous known disease, injury, or surgical intervention involving the brain or central nervous system.
* Moderate or greater hearing loss.
* Presence of a cochlear implant.
* Diagnosed vestibular dysfunction.
* Eye surgery within the previous three months.
* Any history of previous ear surgery.
* Active ear infections or a perforated tympanic membrane.
* Presence of a serious or unstable medical or psychological condition which, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesco Rogers, MD, Study Director — Scion NeuroStim
Locations (1):
- UNC Highgate Specialty Center - UNC Diabetes Care Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caloric Vestibular Stimulation (CVS)
Started | 6
Completed | 0
Not Completed | 6
Not completed — Poor enrollment | 6

BASELINE CHARACTERISTICS:
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/gender was not collected for this study.
  Participants
    Sex/Gender was not collected | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Glycosylated Hemoglobin (A1c)
Description: At the end of the 84 day period of device use, the patient's A1c value will be compared with the baseline value to assess any reduction.
Time Frame: after 84 days of device use
Population: Outcome data was not collected on any patient prior to the study termination.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 0

2. Secondary Outcome: Measurement of Lipid Panel
Description: At the end of treatment (84 day) period, the patient's fasting lipid panel will be taken and compared with the baseline panel to assess any difference in lipid metabolism.
Time Frame: after 84 days of device use
Population: Outcome data was not collected on any patient prior to the study termination.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 0

3. Secondary Outcome: Assessment of Quality of Life
Description: At the end of the 84 day period of device use, the patient's reports on quality of life measures will be compared with baseline values to assess any improvement.
Time Frame: after 84 days of device use
Population: Outcome data was not collected on any patient prior to the study termination.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 0

4. Secondary Outcome: Assessment of Mood
Description: At the end of the 84 day period of device use, the patient's reports on mood measures will be compared with baseline values to assess any improvement.
Time Frame: after 84 days of device use
Population: Outcome data was not collected on any patient prior to the study termination.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 0

5. Secondary Outcome: Assessment of Diabetes Related Self Care
Description: At the end of the 84 day period of device use, the patient's reports on diabetes related self care will be compared with baseline values to assess any improvement.
Time Frame: after 84 days of device use
Population: Outcome data was not collected on any patient prior to the study termination.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 0

6. Secondary Outcome: Feasibility of the Device as an Intervention for the Diabetes Population
Description: At the end of the 84 day period of device use, the patient will be asked to assess the device use experience and note any shortcomings, challenges or difficulties.
Time Frame: after 84 days of device use
Population: Study was halted before any of the participants could complete any of the other endpoints making it impossible to assess the feasibility of the device's use in this population. Data was not collected.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Caloric Vestibular Stimulation (CVS)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
The study was terminated early due to poor enrollment before any of the participants could complete the end of treatment assessments and outcome results could be collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No